CLINICAL TRIAL: NCT05305729
Title: Metabolic FingerPrinting
Acronym: MetaPrint
Status: Recruiting | Type: Observational
Sponsor: Arcensus GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: MetaPrint-2021
Record Dates: First submitted 2022-03-21; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Genetic Disease
Keywords: Metabolic Fingerprint
MeSH Terms: conditions — Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected from all participants.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects with a genetic disease
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The MetaPrint study aims to characterize the metabolic fingerprint of genetic diseases in order to enhance knowledge on the physiological disease status and establish so new tools for diagnosing, monitoring and personalizing treatment of genetic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent is obtained from the participant or from the parent/ legal guardian
* The participant is 2 months or older
* The participant is diagnosed with a genetic disease
* The participant is a first degree relative of a subject diagnosed with a genetic disease

Exclusion Criteria:

* Informed consent is not obtained from the participant or from the parent/ legal guardian
* The participant is younger than 2 months
* The participant is not diagnosed with a genetic disease
* The participant is not a first degree relative of a subject diagnosed with a genetic disease

Min Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All subjects with a confirmed genetic disease as well as their first degree family members can participate in the study.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of newly identified, disease-specific Metabolic Fingerprints | 5 years
  Plasma-derived metabolite profiles that are specific for a particular genetic disease in comparison to healthy controls and other genetic diseases

CONTACTS AND LOCATIONS:
Locations (5):
- University Hospital Center Mother Teresa, Tirana, Albania
- Pakistan (4):
  - The Children's hospital & Institute of child health, Lahore, Punjab Province
  - Pakistan Institute of Medical Sciences (PIMS), Islamabad
  - Children's Hospital & The Institute of Child Health, Multan
  - Khyber institute of Child Health and Children Hospital (KICH), Peshawar

IPD SHARING:
Plan to Share IPD: Undecided
Sharing of IPDs can be discussed after receiving scientific requests.